CLINICAL TRIAL: NCT04997811
Title: Evaluation of Haematological Improvement in Patients With Low-risk MDS by Comparing VBaP With Danazol in Patients Who Have Either Received Erythropoiesis Stimulating Agents (ESA) and Lost Response, Not Responded to ESA or Are Deemed Unlikely to Respond to ESA
Brief Title: Repurposed Drugs to Improve Haematological Responses in Myelodysplastic Syndromes
Acronym: REPAIR-MDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Janet Dunn (Other)
Collaborators: Blood Cancer UK (Unknown); Dudley Group NHS Foundation Trust (Other); University of Birmingham (Other); University of Manchester (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor-Investigator, Prof. Janet Dunn, Professor of Clinical Trials, University of Warwick
Organization: University of Warwick (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOC.11/20-21; 2020-005446-42 (EudraCT Number)
Record Dates: First submitted 2021-07-23; First posted 2021-08-10 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Valproic Acid; Bezafibrate; Medroxyprogesterone; Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VBaP (Experimental): Combination of sodium valproate, bezafibrate, medroxyprogesterone
  Interventions: Drug: Sodium Valproate, Bezafibrate, Medroxyprogesterone
- Danzol (Experimental): Single agent
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Sodium Valproate, Bezafibrate, Medroxyprogesterone — Sodium valproate tablet 1 x 500mg bd, (starting 1 x 200mg bd) Bezafibrate standard release tablet 2 x 200mg tds, (starting 1 x 200mg tds) Medroxyprogesterone acetate tablet 1 x 400mg bd (starting 1 x 400mg od)
  Arms: VBaP
Drug: Danazol — Danazol 1 x 200mg capsules tds, (starting 1 x 200mg od)
  Arms: Danzol

SUMMARY:
Over 7,000 people in the UK are living with Myelodysplastic Syndromes (MDS). Approximately 1,600 of these individuals (23%) die each year from their disease. MDS affects the production of blood cells by the bone marrow, causing chronic fatigue, bleeding, and recurrent infections. Many patients die because their disease transforms into acute myeloid leukaemia (AML) an even more aggressive blood cancer. The general outlook for AML is poor, but when AML arises from MDS it is worse.

REPAIR-MDS seeks to repurpose existing drugs in order to dramatically improve the outlook, health and quality of life of people with MDS. The trial treatments aim to improve the production of healthy functioning blood and immune cells that will fight against infections and boost the immune system's action against the MDS clone.

REPAIR-MDS design is a is a multicentre open label phase 2 randomised controlled trial which will compare VBaP (sodium valproate, bezafibrate, medroxyprogesterone) with danazol in patients who have received either Erythropoiesis Stimulating Agents (ESAs) and lost response, not responded to ESAs or are deemed unlikely to respond to ESAs.

ELIGIBILITY:
Inclusion Criteria (for Randomisation):

1. Provision of written informed consent
2. Age ≥ 18 years and able to give informed consent
3. Diagnosis of Myelodysplastic Syndrome with an IPSS-R score of less than or equal to 3.51
4. Haematological parameters:

   1. Mean haemoglobin < 100 g/l over 16 weeks (pre transfusion) OR
   2. Mean platelets < 100 x 109/l over 16 weeks + evidence of bleeding (assessed using the ISTH Bleeding Assessment Tool) OR
   3. Mean neutrophils < 1.0 x 109/l over 16 weeks + history of infection (the requirement for antimicrobial therapy and hospital admissions associated with infection)
5. No response to Erythroid Stimulating Agents (ESAs) OR Have Ceased to respond to ESAs OR are predicated not to respond to ESAs by current UK guidelines2,3￼ (NB Patients with thrombocytopenia and/or neutropenia, without anaemia, are eligible as they are predicated not to respond to ESAs).
6. ECOG performance status 0-3
7. Expected survival > 12months

Exclusion Criteria (For Randomisation):

Abnormal liver function (if patient has Gilbert's syndrome, then abnormal direct Bilirubin is an exclusion) 2. Cockcroft Gault CrCl < 20ml/min 3. Current systemic treatment for low risk MDS 4. History of Allogeneic Bone Marrow Transplant 5. History of having received ESAs and/or G-CSF in the past 16 weeks 6. Currently receiving statin medication for Secondary Prophylaxis of Cardiovascular Disease, Cerebrovascular Disease or Peripheral Vascular Disease (Please note patients receiving statin medication for Primary Prophylaxis of Cardiovascular Disease - i.e. the patient has no prior history of Ischaemic Heart Disease nor Cerebrovascular Disease - can still be entered, please see section 1.4 Statin use) 7. Currently receiving fibrate medications 8. Currently receiving sodium valproate, carbamazepine or phenytoin for treatment of epilepsy 9. Prior cytotoxic chemotherapy or hypomethylating agents for AML/MDS (eg Azacitidine) 10. Concurrent active malignancy requiring treatment 11. History of any Androgen Dependent Tumour (patients with Prostate Cancer are Excluded when a biopsy proven diagnosis of Prostate Cancer has been made OR their PSA is known to be elevated OR they are on active treatment for Prostate Cancer, including hormonal therapy).

12. Currently receiving Vitamin K-Antagonist Anticoagulation (though patients receiving DOACs (direct oral anticoagulants) can be included) 13. History of Venous Thrombo-Embolism (VTE) 14. Cardiac Failure NYHA Class III or IV 15. Women of childbearing potential, pregnant or lactating 16. The physician or patient consider VBaP or danazol to be inappropriate for the patient 17. Known HIV 18. Abnormally high CK level 19. Presence of isolated del 5q 20. Acute Porphyria 21. Contraindications to any of the trial medications or known hypersensitivity to any of the investigational products (see Appendix C for contraindications) 22. Previous randomisation in the REPAIR-MDS trial 23. Participation in a clinical trial of an investigational medicinal product in the last 16 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Haematological improvement (HI) in each arm and in the trial overall, with 25% or more of the participants having HI in each arm and overall. | 12 months
  HI will be assessed in each participant by comparing post randomisation FBC parameters (Haemoglobin, platelet and neutrophil counts) and transfusion requirements, with their individual baseline as determined by the IWG 2018 haematology response criteria in patients with MDS.

SECONDARY OUTCOMES:
Reduced burden of red cell and/or platelet transfusion in each arm and in the trial overall, as per the IWG 2018 response criteria. | 12 months
  Changes in transfusion requirements will be assessed in each participant by comparison with their individual 16-week lead-in baseline as determined by the IWG 2018 haematology response criteria in patients with MDS.
Duration of haematological response | 12 months
  Clinically meaningful haematological responses that persist for 16 weeks or longer.
Reported improved Health Related Quality of Life scores in each arm and in the trial overall. | 12 months
  The four Health Related Quality of Life questions measure 1) self-perceived health (excellent, very good, good, fair, or poor), (2) number of days out of the past 30 that physical health was not good, (3) number of days out of the past 30 that mental health was not good, and (4) number of days out of the past 30 that usual activities were limited by poor physical or mental health of life scores will be evaluated using established protocols.
Overall survival | Through study completion, an average of 1 year
  Overall survival at close of trial will be reported separately for each trial arm

CONTACTS AND LOCATIONS:
Locations (19):
- United Kingdom (19):
  - Heartlands Hospital, Birmingham, Bordesley Green East
  - Royal Cornwall Hospital NHS Trust, Truro, Cornwall
  - University Hospitals Dorset NHS Foundation Trust, Poole, Dorset
  - Russells Hall Hospital, Dudley, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Broomfield Hospital, Chelmsford, Essex
  - Colchester General Hospital, Colchester, Essex
  - Basingstoke and North Hampshire Hospital,, Basingstoke, Hampshire
  - Royal Hampshire County Hospital, Hampshire Hospitals NHS Foundation Trust, Winchester, Hampshire
  - East Kent Hospitals University Foundation Trust, Canterbury, Kent
  - James Paget University Hospitals NHS Foundation Trust, Gorleston-on-Sea, Norfolk
  - Nottingham City Hospital, Nottingham University Hospitals NHS Trust, Hucknall Road, Nottingham, Nottinghamshire
  - Grampian Health Board, Aberdeen, Scotland
  - Good Hope Hospital, Birmingham, Sutton Coldfield
  - Hull University Teaching Hospitals, Hull
  - Leicester Royal Infirmary, University Hospitals of Leicester NHS Trust, Leicester
  - James Cook University Hospital, South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Royal Gwent Hospital, Aneurin Bevan University Health Board, Newport

REFERENCES:
- See also: REPAIR-MDS Trial Website — http://warwick.ac.uk/fac/sci/med/research/ctu/trials/repairmds